CLINICAL TRIAL: NCT00736671
Title: Striatal and Extra-striatal Mechanisms of Falling in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Nicolaas Bohnen, MD, PhD, Principal Investigator, University of Michigan
Other Study IDs: HUM00003450
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Observational Parkinson's Disease: Observational study of subjects with Parkinson disease
- Observational Normal Control aubjects: Observational study of normal control subjects

SUMMARY:
This research study will evaluate functions of memory, thinking, eye movements and walking and how these relate to the measurement of certain chemicals (acetylcholine and dopamine) in the brain using an imaging procedure called positron emission tomography (PET). You may know that the brain chemical dopamine, a "neurotransmitter" substance (a chemical messenger that nerve cells need to communicate with each other), is important for the brain to control movements and that the brain chemical acetylcholine may have functions related to mental concentration and attention. At the present time, the investigators have no clear information how these two chemicals in the brain of patients with Parkinson's disease are related to the risk of falling.

DETAILED DESCRIPTION:
Although most research in PD has a focus on presynaptic dopaminergic denervation, new lessons may be learned by exploring to what extent alterations in non-motor and non-dopaminergic systems may play a role in the balance impairment in this disorder. This project is designed to evaluate striatal pre-synaptic dopaminergic, cortical, thalamic, and brainstem cholinergic, cognitive, and oculomotor mechanisms underlying the risk of falling and imbalance in PD. The proposed study will exploit advances in our center in the development of dynamic biomathematical modeling of electronic platform data, application of specialized cognitive and oculomotor assessments, and positron emission tomography (PET). This novel multi-system approach holds promise for understanding mechanisms of falling in PD beyond pre-synaptic dopaminergic nigrostriatal denervation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects considered for inclusion will be female or male subjects either currently enrolled or eligible for care at the VA aged 50-85 years, or community volunteers.
* The racial, gender and ethnic characteristics of the proposed subjects population reflect the demographics of the patient population of the VA. However, extra efforts will be made to recruit women and minorities (see table 5).
* Children will be excluded from the study.
* No exclusion criteria shall be based on race, ethnicity, gender, or asymptomatic HIV status.

Exclusion Criteria:

* Inability to stand or walk independently (i.e., patients in Hoehn and Yahr stage IV and V).
* Vertiginous disorder.
* Orthostatic hypotension or unstable cardiovascular disease at risk of syncope (drop in systolic blood pressure of > 20 mm Hg upon standing).
* History of stroke with focal cortical lesions.
* Cerebellar, myelopathic or significant radiculopathy syndrome.
* Diminished light perception in both eyes (< 20/40 corrected OU).
* Intracranial surgery.
* Subjects who have participated in other research protocols such that their cumulative radiation absorbed dose to whole body, gonads, bone marrow or lens of the eye would exceed 5 Rem, or dose to other body organs is more than 15 Rem in preceding 12 months.
* Pregnancy (beta-HCG test within 48 hours of PET study) or breastfeeding.
* Contra-indications to MRI.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease and normal control persons between the ages of 50-85 years are eligible to participate in this study. Participants should be willing and able to comply with study requirements. Normal control persons should not have a history of brain or mental disorders. Both males and females are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2006-07; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Bohnen, Principal Investigator — VAAAHS
Locations (1):
- University of Michigan Functional Neuroimaging, Cognnitive and Mobility Laboratory, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No